CLINICAL TRIAL: NCT03335137
Title: Determining Drug Levels of Beta-lactam Antibiotics in Severe Burned Patients
Acronym: MSBV
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Medical Clinic III (Unknown); Dezernat Apotheke (Unknown)
Responsible Party: Principal Investigator, Tobias Kisch, Principal Investigator, University Hospital Schleswig-Holstein
Other Study IDs: 13-275
Record Dates: First submitted 2017-10-24; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Antibiotics; Severe Burn; Intensive Care
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples are used to determine drug levels of Piperacillin/Tazobactam
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU Patients with Severe Burns: Patients suffering from severe burns treated on a burn unit - Drug Level Monitoring Piperacillin/Tazobactam
  Interventions: Diagnostic Test: Drug Level Monitoring
- ICU Patients without Burns - Drug Level Monitoring: Patient suffering from disease treated on an ICU - Drug Level Monitoring Piperacillin/Tazobactam
  Interventions: Diagnostic Test: Drug Level Monitoring

INTERVENTIONS:
Diagnostic Test: Drug Level Monitoring — Free (unbound) drug concentration 1 hour, 4 hours and 7.5 hours after primary load of piperacillin/tazobactam on day 1 and day 3 after admission

SUMMARY:
At antibiotic stewardship of the University Hospital of Schleswig-Holsten it was noticed that there are much less studies measuring drug levels in severe burned patients than are required. Especially, severe burned patient developing a capillary leak might show lower drug levels than patients without a capillary leak. To compare drug levels of beta-lactam antibiotics, it is the aim of this study to measure pharmacokinetics of Piperacillin/Tazobactam in ICU patients with and without severe burns.

ELIGIBILITY:
Inclusion Criteria:

General

* Adult
* Receiving beta-lactam antibiotic Piperacillin/Tazobactam
* Antibiotic therapy of 3 or more days
* Given informed consent Group 1
* Severe Burn Group 2
* No Severe Burn

Exclusion Criteria:

* Already in another Study
* No useful blood sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated on ICU, in group 1 suffering from severe burns, in group 2 without burns
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Free (unbound) drug concentration 1 hour, 4 hours and 7.5 hours after primary load of piperacillin/tazobactam on day 1 and day 3 after admission | 1 hour, 4 hours and 7.5 hours after primary load of piperacillin/tazobactam on day 1 and day 3 after admission
  Free (unbound) drug concentration 1 hour, 4 hours and 7.5 hours after primary load of piperacillin/tazobactam on day 1 and day 3 after admission

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mailänder, PhD, Study Director — Plastic and Reconstructive Surgery, Hand Surgery, Burn Unit; Walter Raasch, PhD, Study Chair — Institute for experimental and clinical pharmacology and toxicology; Tobias Kisch, MD, Principal Investigator — Plastic and Reconstructive Surgery, Hand Surgery, Burn Unit
Locations (1):
- University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafla K, Tredget EE. Infection control in the burn unit. Burns. 2011 Feb;37(1):5-15. doi: 10.1016/j.burns.2009.06.198. Epub 2010 Jun 18. PMID 20561750
- [Background] Roberts JA. Using PK/PD to optimize antibiotic dosing for critically ill patients. Curr Pharm Biotechnol. 2011 Dec;12(12):2070-9. doi: 10.2174/138920111798808329. PMID 21554211
- [Background] Blanchet B, Jullien V, Vinsonneau C, Tod M. Influence of burns on pharmacokinetics and pharmacodynamics of drugs used in the care of burn patients. Clin Pharmacokinet. 2008;47(10):635-54. doi: 10.2165/00003088-200847100-00002. PMID 18783295
- [Background] Patel BM, Paratz J, See NC, Muller MJ, Rudd M, Paterson D, Briscoe SE, Ungerer J, McWhinney BC, Lipman J, Roberts JA. Therapeutic drug monitoring of beta-lactam antibiotics in burns patients--a one-year prospective study. Ther Drug Monit. 2012 Apr;34(2):160-4. doi: 10.1097/FTD.0b013e31824981a6. PMID 22406650
- [Derived] Olbrisch K, Kisch T, Thern J, Kramme E, Rupp J, Graf T, Wicha SG, Mailander P, Raasch W. After standard dosage of piperacillin plasma concentrations of drug are subtherapeutic in burn patients. Naunyn Schmiedebergs Arch Pharmacol. 2019 Feb;392(2):229-241. doi: 10.1007/s00210-018-1573-6. Epub 2018 Oct 27. PMID 30368548